CLINICAL TRIAL: NCT05465850
Title: Shade Matching Potential of Universal Shade Resin Composite Materials Compared to Multi Shade Resin Composite in Restoration of Carious Cervical Lesions in Anterior Teeth ( Randomized Clinical Trial ) - 1 Year Follow up
Brief Title: Shade Matching Potential of Universal Shade Resin Composite Materials Compared to Multi Shade Resin Composite in Restoration of Carious Cervical Lesions in Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Khaled Mokhtar Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019428237
Record Dates: First submitted 2022-06-27; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Class V Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Filtek Z350XT (Active Comparator)
  Interventions: Diagnostic Test: Modified USPHS criteria
- Essentia universal shade, GC composite (Experimental)
  Interventions: Diagnostic Test: Modified USPHS criteria
- Omnichroma composite (Experimental)
  Interventions: Diagnostic Test: Modified USPHS criteria

INTERVENTIONS:
Diagnostic Test: Modified USPHS criteria — It assess the restorations with visual inspection using a mirror and explorer. It includes Marginal integrity, shade matching, retention, marginal discoloration, gingival inflammation, and recurrent caries.

SUMMARY:
The aim of the study is to clinically evaluate the shade matching and clinical performance of the Universal shade composites Omnichroma and GC Essentia versus the multi shade composite Filtek Z350XT in restoring cervical lesions of anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Class V carious lesions in anterior teeth
* Vital upper or lower anterior teeth with no signs of irreversible pulpitis and necrosis.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth

Exclusion Criteria:

* Deep carious defects ( Close to pulp, less than 1 mm distance)
* Periapical pathology or signs of pulpal pathology
* Endodontically treated teeth
* Tooth hypersensitivity
* Possible prosthodontic restoration of teeth
* Heavy occlusion and occlusal contacts or history of bruxism
* Severe periodontal affection
* Lesions in premolars and molars
* Posterior teeth

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Clinical performance (USPHS criteria) | baseline: 1 week
  USPHS criteria
Clinical performance (USPHS criteria) | 6 months
  USPHS criteria
Clinical performance (USPHS criteria) | 12 months
  USPHS criteria

IPD SHARING:
Plan to Share IPD: No